CLINICAL TRIAL: NCT03317405
Title: Phase I Trial of Endoxifen Gel Versus Placebo Gel in Women Undergoing Breast Surgery
Brief Title: Phase I Trial of Endoxifen Gel Versus Placebo in Women Undergoing Breast Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2017-01921; NCI-2017-01921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI2017-09-01 (Other: Northwestern University); NWU2017-09-01 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2017-10-20; First posted 2017-10-23 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Ductal Carcinoma In Situ; Breast Lobular Carcinoma In Situ; Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (endoxifen hydrochloride) (Experimental): Participants apply endoxifen hydrochloride gel to both breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Interventions: Drug: Endoxifen Hydrochloride; Other: Questionnaire Administration
- Cohort II (placebo) (Placebo Comparator): Participants apply placebo to both breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Interventions: Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Endoxifen Hydrochloride — Apply to the skin
  Other Names: Z-Endoxifen HCl; Z-Endoxifen Hydrochloride
  Arms: Cohort I (endoxifen hydrochloride)
Other: Placebo Administration — Apply to the skin
  Arms: Cohort II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase I trial studies the side effects and best dose of endoxifen hydrochloride in treating participants who are undergoing breast surgery. Endoxifen hydrochloride may treat or reduce the risk of breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the dermal tolerability and safety of endoxifen hydrochloride (endoxifen [ENX]) gel administered topically to both breasts at two doses: 10 mg daily (5 mg per breast) and 20 mg daily (10 mg per breast) in comparison to vehicle placebo gel, using objective assessments based on Common Terminology Criteria for Adverse Events (CTCAE) criteria.

SECONDARY OBJECTIVES:

I. To measure the breast tissue concentrations of (E) and (Z) isomers of N-desmethyl-4-hydroxytamoxifen (ENX) and 4-hydroxytamoxifen (4-OHT) at each dose (10 mg per day and 20 mg per day).

II. To measure the plasma concentrations of (E) and (Z) isomers ENX and 4-OHT at each dose (10 mg per day and 20 mg per day).

III. To measure serum estrogenic response to topical ENX gel therapy in comparison to vehicle placebo gel (sex hormone binding globulin and insulin-like growth factor [IGF] pathway proteins).

IV. To assess changes in coagulation parameters (factor VIII, factor IX, vWF, protein S) in response to ENX gel therapy in comparison to vehicle placebo gel.

V. To assess symptoms related to use of endoxifen gel in comparison to vehicle placebo gel, as assessed by the Breast Cancer Prevention Trial (BCPT) Eight Symptom Scale (BESS) questionnaire.

EXPLORATORY OBJECTIVE:

I. Using pathological lesion-matched pre- and post-therapy tissue samples, to explore the potential therapeutic effects of the two doses of ENX gel in comparison to vehicle placebo gel: a) by IHC, Ki67 labelling (for cell proliferation), estrogen receptor (ER), progesterone receptor (PR) expression (for estrogen blockade); b) by expression of a panel of genes reported to change with ENX exposure (using nanostring assays).

OUTLINE: Participants are randomized in Cohorts 1 and 2. All subjects in Cohort 3 will receive active agent.

COHORT I: Participants apply endoxifen hydrochloride gel to both breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.

COHORT II: Participants apply placebo to both breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.

COHORT III: Participants apply endoxifen hydrochloride gel to both breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.

After completion of study treatment, participants are followed up at 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for unilateral or bilateral mastectomy for breast cancer therapy, pathology confirmed stage 0-III (including ductal carcinoma in situ), or prophylaxis (BRCA1/2 mutation carriers, women with strong family history or lobular carcinoma in situ or other conditions where prophylactic mastectomy has been elected)
* Age >= 18 years (since breast cancer is not a pediatric disease and no safety data are available for ENX use in children)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Total bilirubin < 1.5 x upper limit of normal (ULN) (in women with prior documented bilirubin elevations consistent with Gilbert's syndrome, total bilirubin up to 3 x ULN will be allowed)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) < 2.5 x ULN
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x ULN
* Creatinine < 2 x ULN
* Alkaline phosphatase < 2.5 x ULN
* Blood urea nitrogen < 2 x ULN
* Ability to understand and the willingness to sign a written informed consent document which includes a requirement to apply study agent to sensitive body parts daily
* Willingness and ability to schedule mastectomy 21-28 days following start of study agent; women with breast implants may participate
* Willingness to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the duration of study agent dosing
* Negative urine or serum pregnancy test result, for participants of child bearing potential; female of child-bearing potential is any woman (regardless of sexual orientation, whether she has undergone a tubal ligation, or remains celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; AND has had a menstrual period at any time in the preceding 12 consecutive months)
* The effects of topical ENX gel on the developing human fetus are unknown; for this reason, women of child-bearing potential and their male partners must agree to use effective forms of birth control (abstinence is not an allowed method) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

Exclusion Criteria:

* The presence of gross skin invasion/ulceration by the breast cancer, or inflammatory changes with skin edema AND erythema; Note: Paget's disease is permitted
* Women receiving a "nipple delay" procedure prior to mastectomy
* Women with skin diseases (psoriasis, eczema)
* A history of thromboembolic disorder
* Endometrial intraepithelial neoplasia (also known as atypical hyperplasia) or a high risk of uterine cancer, defined here as known carriers of Lynch syndrome mutations (MLH1, MSH2, MSH6, PMS2)
* Participants may not have received any other investigational agents in the previous 3 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tamoxifen
* Taken tamoxifen or other selective estrogen/progesterone receptor modulators (SERMs/SPRMs) within two years prior to entering study or been required to discontinue SERM therapy due to thromboembolic or uterine toxicity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of prior breast cancer-specific therapy within the previous 2 years (chemotherapy, radiation, anti-HER2 agents, endocrine agents, everolimus, CDK4-6 inhibitors); previous unilateral radiation of the contralateral side in women scheduled for mastectomy is allowed; study gel will be applied to both breasts
* History of prior mastectomy
* Pregnant or breastfeeding
* Patients receiving neoadjuvant chemotherapy with curative intent
* Men are excluded from this study since breast cancer is men is rare and there are no data regarding skin penetration of topical breast cancer prevention agents through male chest wall skin (which is thicker and harrier than female chest wall skin)
* Current users of other topical medications on the breast skin must be willing and able to discontinue use for the duration of participation; body lotion and other non-medicinal topical compounds may be applied > 4 hours after study gel application

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2026-08-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Seema A Khan, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Endoxifen Hydrochloride Gel 10 mg Daily: Participants apply endoxifen hydrochloride gel 5 mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 5 mg: Apply to each breast daily for total dose of 10 mg daily
  Questionnaire Administration: Ancillary studies
- Endoxifen Hydrochloride Gel 20 mg Daily: Participants apply endoxifen hydrochloride gel 10 mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 10 mg: Apply to each breast daily for total dose of 20 mg daily
  Questionnaire Administration: Ancillary studies
- Placebo: Participants apply placebo to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Placebo Administration: Apply to each breast daily
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg Daily | Placebo
Started | 16 | 8 | 8
Completed | 15 | 7 | 7
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Surgery Rescheduled | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Women who are scheduled for mastectomy, either for risk reduction, or for breast cancer or DCIS therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg Daily | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 8 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 8 | 32
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 13 | 7 | 7 | 27
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 11 | 6 | 5 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dermal Toxicity on Breast Skin at the Application Site
Description: Number of participants with dermal toxicity on breast skin at the transdermal gel application site. Will be assessed by Common Terminology Criteria for Adverse Events version 4.
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Groups:
- Endoxifen Hydrochloride Gel 10 mg Daily: Participants apply endoxifen hydrochloride gel 5 mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 5 mg: Apply to each breast daily for total dose of 10 mg daily
- Endoxifen Hydrochloride Gel 20 mg Daily: Participants apply endoxifen hydrochloride gel 10mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 10 mg: Apply to each breast daily for total dose of 20 mg daily
- Placebo: Participants apply placebo to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Placebo Administration: Apply to each breast daily
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg Daily | Placebo
Number analyzed (Participants) | 16 | 8 | 8
Participants | 4 | 2 | 0

2. Secondary Outcome: Drug Concentration in Tissue
Description: Concentrations of (E) and (Z) Isomers ENX in right and left breast tissue at end of intervention (up to 4 weeks) in tissue samples
Time Frame: up to 28 days
Population: Participants with right and/or left breast tissue samples pre- and post-therapy
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg Daily | Placebo
Number analyzed (Participants) | 15 | 5 | 6
ng/g
  Central Subareolar Left Breast Z_ENX: number analyzed (Participants) | 15 | 4 | 6
  Central Subareolar Left Breast Z_ENX | 0.47 [0.15 to 0.79] | 0.76 [0.65 to 1.01] | 0.00 [0.00 to 0.00]
  Central Subareolar Left Breast E_ENX: number analyzed (Participants) | 15 | 4 | 6
  Central Subareolar Left Breast E_ENX | 0.16 [0.16 to 0.28] | 0.25 [0.16 to 0.39] | 0.00 [0.00 to 0.00]
  Central Subareolar Right Breast Z_ENX: number analyzed (Participants) | 12 | 4 | 3
  Central Subareolar Right Breast Z_ENX | 0.37 [0.15 to 0.44] | 1.00 [0.62 to 1.51] | 0.00 [0.00 to 0.00]
  Central Subareolar Right Breast E_ENX: number analyzed (Participants) | 12 | 4 | 3
  Central Subareolar Right Breast E_ENX | 0.16 [0.16 to 0.16] | 0.30 [0.16 to 0.58] | 0.00 [0.00 to 0.08]
  Central Deepest Left Breast Z_ENX: number analyzed (Participants) | 15 | 4 | 5
  Central Deepest Left Breast Z_ENX | 0.40 [0.15 to 1.73] | 1.55 [0.34 to 2.85] | 0.00 [0.00 to 0.00]
  Central Deepest Left Breast E_ENX: number analyzed (Participants) | 15 | 4 | 5
  Central Deepest Left Breast E_ENX | 0.16 [0.16 to 1.39] | 0.91 [0.16 to 1.78] | 0.00 [0.00 to 0.16]
  Central Deepest Right Breast Z_ENX: number analyzed (Participants) | 12 | 4 | 3
  Central Deepest Right Breast Z_ENX | 0.46 [0.15 to 1.58] | 2.57 [1.3 to 15.06] | 0.00 [0.00 to 0.100]
  Central Deepest Right Breast E_ENX: number analyzed (Participants) | 12 | 4 | 3
  Central Deepest Right Breast E_ENX | 0.28 [0.16 to 1.69] | 1.70 [1.13 to 17.20] | 0.00 [0.00 to 0.00]
  Lateral Surface Left Breast Z_ENX: number analyzed (Participants) | 15 | 4 | 6
  Lateral Surface Left Breast Z_ENX | 0.34 [0.15 to 0.75] | 0.81 [0.58 to 1.00] | 0.00 [0.00 to 0.00]
  Lateral Surface Left Breast E_ENX: number analyzed (Participants) | 15 | 4 | 6
  Lateral Surface Left Breast E_ENX | 0.16 [0.16 to 0.50] | 0.27 [0.16 to 0.42] | 0.00 [0.00 to 0.00]
  Lateral Surface Right Breast Z_ENX: number analyzed (Participants) | 11 | 5 | 3
  Lateral Surface Right Breast Z_ENX | 0.45 [0.15 to 1.38] | 1.20 [0.99 to 1.27] | 0.00 [0.00 to 0.08]
  Lateral Surface Right Breast E_ENX: number analyzed (Participants) | 11 | 5 | 3
  Lateral Surface Right Breast E_ENX | 0.16 [0.16 to 1.12] | 0.39 [0.16 to 0.47] | 0.00 [0.00 to 0.00]

3. Secondary Outcome: Drug Concentration in Plasma
Description: Concentration of (E) and (Z) Isomers ENX in plasma at the end of intervention (up to 4 weeks)
Time Frame: baseline and up to 28 days
Population: Protocol adherent participants (took minimum 80% of the required doses based on diary record and the remaining gel weight) with plasma samples pre- and post-therapy
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Endoxifen Hydrochloride Gel 10 mg: Participants apply endoxifen hydrochloride gel 5 mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 5 mg: Apply to each breast daily for total dose of 10 mg daily
- Endoxifen Hydrochloride Gel 20 mg: Participants apply endoxifen hydrochloride gel 10 mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 10 mg: Apply to each breast daily for total dose of 20 mg daily
- Placebo: Participants apply placebo to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Placebo Administration: Apply to each breast skin
Arm/Group | Endoxifen Hydrochloride Gel 10 mg | Endoxifen Hydrochloride Gel 20 mg | Placebo
Number analyzed (Participants) | 15 | 5 | 7
ng/ml
  Z_ENX | 0.15 [0.15 to 0.15] | 0.44 [0.15 to 0.54] | 0.00 [0.00 to 0.00]
  E_ENX | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

4. Secondary Outcome: Change in Plasma Estrogenic and Coagulation Parameters
Description: Change in plasma Estrogenic and Coagulation Parameters from baseline to end of intervention (up to 28 days) including: IGF1, IGFBP3, SHBG.
Time Frame: baseline and up to 28 days
Population: Participants with plasma samples pre- and post-therapy
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg | Placebo
Number analyzed (Participants) | 15 | 6 | 7
ng/ml
  IGF1 | -1.7 [-9.9 to 6.6] | 3.0 [-8.6 to 15] | -1.0 [-17 to 15]
  IGFBP3 | 48 [-29 to 125] | -2.5 [-216 to 211] | -60 [-205 to 84]
  SHBG | -9.4 [-26 to 6.8] | 1.9 [-13 to 17] | -4.4 [-12 to 3.8]

5. Secondary Outcome: Change in Pre-therapy and Post-therapy Symptoms Captured by BESS Questionnaire
Description: Assessed using the Breast Cancer Prevention Trial (BCPT) Eight Symptom Scale (BESS) questionnaire. A patient reported outcome, subscale scores range from 0 (Not at All) to 4 (Extremely) when asked about experiencing symptoms. A positive change in scores indicates an increase in symptoms experienced and a negative change in scores indicates a decrease in symptoms experienced.
Time Frame: baseline and up to 60 days
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Groups:
- Endoxifen Hydrochloride Gel 20 mg Daily: Participants apply endoxifen hydrochloride gel 10 mg to each breast skin and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 10 mg: Apply to each breast daily for total dose of 20 mg daily
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg Daily | Placebo
Number analyzed (Participants) | 15 | 7 | 7
change in score on a scale
  Cognitive | -0.16 [-0.60 to 0.29] | -0.05 [-1.0 to 0.88] | -0.19 [-0.62 to 0.24]
  Body Pain | -0.18 [-0.44 to 0.08] | -0.38 [-1.2 to 0.48] | -0.10 [-0.73 to 0.54]
  Vasomotor | -0.02 [-0.26 to 0.21] | -0.05 [-0.16 to 0.07] | 0.19 [-0.64 to 1.0]
  Gastrointestinal | -0.07 [-0.19 to 0.06] | -0.24 [-0.53 to 0.06] | 0.10 [-0.20 to 0.39]
  Sexual Problems | 0.13 [-0.15 to 0.42] | -0.57 [-1.8 to 0.64] | -0.29 [-0.74 to 0.17]
  Body Image | -0.20 [-0.54 to 0.14] | -0.64 [-1.3 to 0.00] | -0.43 [-1.4 to 0.55]
  Vaginal | 0.13 [-0.21 to 0.47] | -0.29 [-0.77 to 0.20] | -0.24 [-0.53 to 0.06]
  Bladder Problem | 0.03 [-0.04 to 0.10] | -0.86 [-1.8 to 0.06] | 0.07 [-0.10 to 0.25]

ADVERSE EVENTS:
Time Frame: AEs collected from the time informed consent was signed and baseline procedures were completed through 60 days post-intervention. In total AEs collected for a period of up to 3 months.
Groups:
- Endoxifen Hydrochloride Gel 10 mg Daily: Participants apply endoxifen hydrochloride gel 5 mg to each breast skin daily and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 5 mg: Apply to each breast daily for total dose of 10 mg daily
  Questionnaire Administration: Ancillary studies
- Endoxifen Hydrochloride Gel 20 mg Daily: Participants apply endoxifen hydrochloride gel 10 mg to each breast skin daily and keep it untouched over at least 4 hours once daily for 21-28 days before breast surgery.
  Endoxifen Hydrochloride 10 mg: Apply to each breast daily for total dose of 20 mg daily
  Questionnaire Administration: Ancillary studies
Arm/Group | Endoxifen Hydrochloride Gel 10 mg Daily | Endoxifen Hydrochloride Gel 20 mg Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/16 | 3/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endoxifen Hydrochloride Gel 10 mg Daily (N=16) | Endoxifen Hydrochloride Gel 20 mg Daily (N=8) | Placebo (N=8)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (7) | 3 (6) | 1 (1) — All events were at the application site and described as: burning, dryness, dry skin, itchy mild rash, itchiness, itchy skin, itchy spots, skin irritation, and soreness.
Hot flashes (Vascular disorders) | 1 (1) | 1 (1) | 3 (5)
Vaginal Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT03317405/Prot_SAP_ICF_001.pdf